CLINICAL TRIAL: NCT07232654
Title: A Clinical Study to Evaluate the Safety and Efficacy of Iparomlimab/Tuvonralimab Injection (QL1706, a Bifunctional Mabpair Product of Anti-PD-1 and Anti-CTLA-4 Antibodies) in Combination With Concurrent Chemoradiotherapy in Patients With Locally Advanced Cervical Cancer
Brief Title: Iparomlimab/Tuvonralimab Injection Plus CCRT in LACC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LING YING WU, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-IIT-CC-001
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: LOCALLY ADVANCED CERVICAL CANCERS
Keywords: QL1706; Concurrent Chemoradiation Therapy; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants will receive 1 cycle of Iparomlimab/Tuvonralimab induction therapy followed by concurrent chemotherapy and radiotherapy. Iparomlimab/Tuvonralimab will be administered by intravenous infusion at a dose of 5 mg/kg on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator or withdraw consent or have completed 2 years of Iparomlimab/Tuvonralimab treatment.
  Interventions: Drug: Iparomlimab/Tuvonralimab; Drug: Cisplatin; Radiation: Brachytherapy and External Beam Radiotherapy
- Arm 2 (Experimental): Participants will receive Iparomlimab/Tuvonralimab combined with concurrent chemotherapy and radiotherapy.
  Iparomlimab/Tuvonralimab will be administered by intravenous infusion at a dose of 5 mg/kg on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator or withdraw consent or have completed 2 years of Iparomlimab/Tuvonralimab treatment.
  Interventions: Drug: Iparomlimab/Tuvonralimab; Drug: Cisplatin; Radiation: Brachytherapy and External Beam Radiotherapy

INTERVENTIONS:
Drug: Iparomlimab/Tuvonralimab — IV infusion
Drug: Cisplatin — IV infusion
Radiation: Brachytherapy and External Beam Radiotherapy — Radiation

SUMMARY:
This study is a clinical study to evaluate the safety and efficacy of Iparomlimab/Tuvonralimab Injection (QL1706, a Bifunctional Mabpair Product of Anti-PD-1 and Anti-CTLA-4 Antibodies) in Combination With Concurrent Chemoradiotherapy in Patients With Locally Advanced Cervical Cancer.

ELIGIBILITY:
Inclusion criteria

* Informed consent.
* Female patients aged ≥18 years and ≤ 75 years at time of inform consent signature
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Expected survival ≥ 3 months
* Patients must have histologically confirmed diagnosis of HPV-related cervical squamous, or adenocarcinoma, or adenosquamous carcinoma
* FIGO 2018 stage T3a-4a (III-IVA), N1 (positive lymph node metastasis on CT/MRI with short-axis ≥1 cm, or PET-CT showing one or more lymph node metastases with SUVmax ≥2.5), M0
* Has at least one evaluable disease per RECIST 1.1
* Has adequate organ function

  * Hematology: ANC ≥1.5 ×10⁹/L; platelets ≥100 ×10⁹/L; hemoglobin ≥90 g/L (no blood transfusion or growth factor support within 7 days)
  * Renal: CrCl ≥50 mL/min (Cockcroft-Gault formula), urine protein <2+ or 24h <1.0 g
  * Hepatic: Total bilirubin ≤1.5×ULN; AST and ALT ≤2.5×ULN
  * Coagulation: INR and APTT ≤1.5×ULN
  * Cardiac: LVEF ≥50%
* Women of childbearing potential: a negative urine or serum pregnancy test within 3 days prior to the first dose of study drug (if the urine pregnancy test result cannot be confirmed as negative, a serum pregnancy test must be performed, and the serum result will be considered definitive).If a female participant of childbearing potential engages in sexual activity with a male partner who is not surgically sterile, she must use an acceptable method of contraception starting from screening and agree to continue using the same contraception for 120 days after the last dose of study drug. Whether to discontinue contraception after this period should be discussed with the investigator
* Willingness to comply with the study procedures before study entry

Main Exclusion Criteria:

* Cervical cancer of other histology (e.g., neuroendocrine carcinoma, sarcoma)
* Evidence of distant metastasis
* Prior total hysterectomy (subtotal or cervical-sparing surgery allowed)
* Unable or unwilling to receive brachytherapy
* Prior treatment with immune checkpoint inhibitors or other tumor immunotherapy
* Systemic corticosteroid (>10 mg/day prednisone or equivalent) or immunosuppressive therapy within 2 weeks (exceptions: inhaled/topical ≤10 mg/day, physiologic replacement ≤10 mg/day, premedication for hypersensitivity).
* Immunomodulatory drugs within 2 weeks (e.g., thymosin, interferons, IL-2)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
2-year PFS rate | up to 24 months

SECONDARY OUTCOMES:
ORR | Up to approximately 24 months
PFS | Up to approximately 24 months
DCR | Up to approximately 24 months
DoR | Up to approximately 24 months
OS | Up to approximately 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Beijing, China